CLINICAL TRIAL: NCT03010605
Title: Evaluation of the Measuring Every Day, Patient Incentive Device, as an Adjunct to Conventional Physical Therapy in the Acceleration of Flexion and Extension Capability in the Post-Operative Total Knee Arthroplasty Patient: A Prospective, Randomized Study
Brief Title: Measuring Every Day (MED) Study
Acronym: MED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Christ Hospital (Other)
Responsible Party: Principal Investigator, Dr. Michael Swank, Principal Investigator, The Christ Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Total Knee Arthroplasty
Keywords: physical therapy post total knee replacement; range of motion; goniometry
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care physical therapy (Active Comparator): Patients will receive 2 weeks of in-home physical therapy consisting of 3 sessions per week followed by 4 weeks of outpatient physical therapy three times weekly.
  Interventions: Other: Physical Therapy
- MED Device (Active Comparator): Patients will perform 10 repetitions with the MED device 3 times daily at 8am, 2pm, and 8pm and will transmit the 10th measurement of each time point to the clinicians office.
  Interventions: Device: Measuring Every Day Device

INTERVENTIONS:
Device: Measuring Every Day Device
  Other Names: MED Device
  Arms: MED Device
Other: Physical Therapy
  Arms: Standard of care physical therapy

SUMMARY:
Achieving adequate range of motion post Total Knee Arthroplasty(TKA) is an important goal for return to optimum function. Traditionally, adequate range of motion has been achieved by a combination of in-home and outpatient physical therapy. While physical therapy is successful, it has the limitation of cost and availability. As copayments rise, patients may decide that they cannot afford physical therapy, potentially compromising the outcome of their surgery and successful return to function.

It is assumed that having an easy and fun to use, patient administered, incentive device that provides accurate, quantitative flexion and extension measurements may accelerate patient mobility and return to function after TKA. The Measuring Every Day (MED) portable goniometer is commercially available and provides objective, consistent range of motion measurements that are recorded and can be sent electronically to the clinician's office potentially enabling earlier clinical or therapy adjustments or modifications to the prescribed therapy.

Goniometry is a commonly used tool to measure and document range of motion (ROM) during clinical evaluation or a physical therapy examination. The technique is used to assess the limitations of a patient's joint and provide information to the clinician that may help determine further treatment.

The study is designed to compare range of motion measurement data for 6 weeks in patients that have been randomized to receive either traditional physical therapy or the MED device. The hypothesis is that patients who use the MED device achieve equivalent range of motion at six weeks as compared to patients participating in traditional standard of care physical therapy.

DETAILED DESCRIPTION:
The MED is a commercially available, digital range of motion monitoring device for patients recovering from knee surgery. It displays both flexion and extension measurements and has the option of connecting to an Apple or Android device to send data to the clinician's office for review. Patients will have the capability to log on to the Measuring Every Day website with an assigned username and a password which they create. This will allow them to view their progress and send messages to the study team. Study team members will also have access to this website for review and the ability to send and receive messages. All shared files will reside on an Amazon HIPAA compliant platform.

This is a prospective, randomized, unblinded, single-center study to compare the MED device to traditional physical therapy. The study will include 46 patients who have undergone successful, unilateral total knee arthroplasty. All patients will receive a minimum of 2 physical therapy sessions prior to hospital discharge and also be instructed to flex and extend their operative knee 10 times every 15 minutes while awake as per standard of care after discharge. Patients will be randomized in a 1:1 ratio prior to discharge from the hospital to either: 1) total knee arthroplasty standard of care rehab which consists of 2 weeks of in-home physical therapy consisting of 3 sessions per week starting within 48 hours of hospital discharge, followed by 4 weeks of out-patient therapy three times weekly, or 2) ten repetitions with the MED device three times daily at 8:00am, 2:00pm and 8:00pm. Patients will transmit the 10th measurement of each time point to the clinician's office. Patients randomized to the MED device will be trained on the use of the device prior to hospital discharge.

All enrolled subjects will return to the surgeon's office at Week 2 to have their index knee range of motion measured by the PI or study coordinators with the MED device. If subjects enrolled in the MED device arm do not have a minimum flexion of 90 degrees and extension of -25 degrees, they will be considered screen failures and return to traditional physical therapy.

All enrolled subjects will return to the surgeon's office at Week 6 to have their index knee range of motion measured by the PI or study coordinators using the MED device with the goal of achieving a minimum flexion of 120 degrees and an extension of 0 degrees.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to provide written informed consent.
2. Age 18 - 64 years of age
3. Subject has undergone successful unilateral total knee arthroplasty for degenerative joint disease
4. Subject has access to an Apple device with Bluetooth capability
5. Subject is able to demonstrate the capability of setting up and using an Apple application for remote data collection and transmission
6. Subject is able to demonstrate capability of correctly using the MED device
7. Subject is able to comply with post-operative visits and evaluations

Exclusion Criteria:

1. Subject is scheduled for an index knee revision surgery
2. Subject has pre-operative flexion range of motion less than 110 degrees
3. Subject has a pre-operative flexion contracture greater than 15 degrees.
4. Subject has additional joint replacement surgery scheduled within the six week study period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Index Knee Flexion of 90 degrees | 2 weeks post-op
Index Knee Extension of -25 degrees | 2 weeks post-op
Index Knee Flexion of 120 degrees | 6 weeks post-op
Index Knee Extension of 0 degrees | 6 weeks post-op

CONTACTS AND LOCATIONS:
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided